CLINICAL TRIAL: NCT04926272
Title: Amyloid-beta PET Imaging With 18F-92 in Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRCTA, ECFAH of FMU [2021]130
Record Dates: First submitted 2021-06-07; First posted 2021-06-15 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-92, PET/CT (Experimental): PET/CT perform after injecting 18F-92
  Interventions: Drug: 18F-92

INTERVENTIONS:
Drug: 18F-92 — Intravenous injection of one dose of 0.10mCi/kg(±5%) 18F-92. Each subject receive a single intravenous injection of 18F-92, and undergo PET/CT imaging within the specificed time.

SUMMARY:
Alzheimer's disease is a neurodegenerative disease. Numerous studies have reported that β-amyloid (Aβ) is an important marker for the diagnosis of AD. 18F-92 molecular probe is a novel molecularly targeted imaging agent, which can rapidly penetrate the blood-brain barrier and has high affinity and selectivity for Aβ protein. In this study, 18F-92 PET/CT was used to monitor the regional distribution and the degree of deposition in patients with Alzheimer's disease, and compared with clinical symptoms (neuropsychometry) to evaluate its application value in the diagnosis of AD.

DETAILED DESCRIPTION:
Healthy volunteers as well as patients meeting Alzheimer's criteria will be recruited for this study.

We will use PET/CT imaging technology to scan each participant's whole body or head and collect image data for analysis to evaluate the distribution and metabolism of 18F-92 in the subject's body. Time from drug injection to scan completion is approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their families complain of significant memory impairment;
* Objective memory impairment (e.g., tests of article identification, recall, delayed memory);
* Meets Alzheimer's criteria for DSMIV and NINCDS-ADRDA;
* Be able to obtain complete diagnosis and treatment records and be able to carry out long-term follow-up;
* Signed written consent.

Exclusion Criteria:

* Nervous system diseases: including brain tumors, craniocerebral trauma, multiple sclerosis, epilepsy, etc.;
* Psychiatric disorders: including anxiety disorder, affective disorder, severe psychosis, or drug-induced psychosis;
* Pregnancy or lactation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
standardized uptake value ratio (SUVR) | From right after tracer injection to 2-hours post-injection
  the ratio of radioactivity in a cerebral region to that in the cerebellum as a reference
Aβ42 in CSF | Within 2 hours prior to tracer injection
  Aβ42 (amyloid beta isoform 42) is significantly lower in the cerebrospinal fluid of patients with Alzheimer's disease and is one of the biomarkers used clinically to diagnose Alzheimer's disease
t-tau in CSF | Within 2 hours prior to tracer injection
  t-tau (total tau) is significantly increased in the cerebrospinal fluid of patients with Alzheimer's disease and is one of the biomarkers used clinically to diagnose Alzheimer's disease
p-tau in CSF | Within 2 hours prior to tracer injection
  p-tau (tau phosphorylated at Thr-181) is significantly increased in the cerebrospinal fluid of patients with Alzheimer's disease and is one of the biomarkers used clinically to diagnose Alzheimer's disease
MMSE (Mini-mental State Examination) | Within 2 hours prior to tracer injection
  The commonly used neuropsychological evaluation scale in clinical practice can comprehensively reflect the intellectual status and the degree of cognitive decline of the subjects. 30 points total, lower scores represent worse cognitive function, normal: 27-30 points; cognitive dysfunction: < 27; mild: 21-26; moderate: 10-20; severe: 0-9
MoCA (Montreal Cognitive Assessment) | Within 2 hours prior to tracer injection
  A scale used clinically for cognitive function screening, with a full score of 30, ≥ 27 being normal, 18-26 being mild cognitive impairment, 10-17 being moderate, and less than 10 being severe

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No